CLINICAL TRIAL: NCT05363865
Title: Digital, Community-Led, Social Action Initiative to Reduce Opioid Vulnerability and HIV/HCV in Rural Areas of the Midwest and Appalachia
Brief Title: Digital Community to Improve Health in Rural Areas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 390234
Record Dates: First submitted 2022-04-21; First posted 2022-05-06 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: HIV Infections; Hepatitis C Virus Infection
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Clusters will be randomized to either the intervention or the standard of care.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be unaware of the experimental condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Community Intervention (Experimental): Participants will participate in an online community with structured sessions as well as the ability to communicate freely with others.
  Interventions: Behavioral: Virtual Community Intervention
- Standard of Care (Active Comparator): Participants will be exposed to what's disseminated within their communities
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Virtual Community Intervention — Modules of community building, HIV/HCV prevention, drug and service stigma, identification of mental health problems
  Arms: Virtual Community Intervention
Behavioral: Standard of Care — health websites and county information provided to participants
  Arms: Standard of Care

SUMMARY:
The study is a cluster randomized controlled trial developed in counties located in Appalachia and the Midwest. We will prioritize counties from states with high risk for HIV and HCV infection associated with injection drug use.

DETAILED DESCRIPTION:
The study will randomize clusters with groups of participants to an intervention or a standard of care condition.

ELIGIBILITY:
Inclusion Criteria:

* Lives in target zip codes
* Half not using illicit substances (not including marijuana) currently or in the past
* Half using illicit substances (not including marijuana) currently or in the past

Exclusion Criteria:

* Under the age of 18
* Not in target zip codes

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Composite of Six Yes/No Behaviors Promoted by Intervention | Baseline, Session 2 [Experimental Condition Only], Immediate Follow-Up (3 Weeks), 3 months, 6 months
  Measures:
  Sum of Yes to (a) self-testing for HIV, (b) self-testing for HCV, (c) HIV prevention, (d) requesting Naloxone, (e) carrying Naloxone, and (f) making at least one social connection (new or reestablished).
  Continuous (0 to 6)

SECONDARY OUTCOMES:
HIV and HCV Testing | Baseline [Control not offered testing at baseline], Session 2 [Experimental Condition Only], Immediate Follow-Up (3 Weeks), 3 months, 6 months
  Measures:
  Test for HIV
  Test for HCV
  Binary (Yes/No)
HIV Prevention Behaviors | Baseline, Session 2 [Experimental Condition Only], Immediate Follow-Up (3 Weeks), 3 months, 6 months
  Measures:
  If they have HIV risk:
  Using PrEP (Pre-Exposure Prophylaxis)
  Binary (Yes/No)
  Use a condom when you had sex
  Continuous (Numeric)
  Use of syringe service programs
  Binary (Yes/No)
  Disinfecting injection equipment
  Binary (Yes/No)
Requesting Naloxone (Narcan) | Baseline[Control not offered Naloxone at baseline], Session 2 [Experimental Condition Only], Immediate Follow-Up (3 Weeks), 3 months, 6 months
  Measures:
  If your state allows it, would you like us to send you Narcan/naloxone?
  Binary (Yes/No)
Carrying Naloxone (Narcan) | Baseline[Control not offered Naloxone at baseline], Session 2 [Experimental Condition Only], Immediate Follow-Up (3 Weeks), 3 months, 6 months
  Measures:
  Carry Naloxone Frequency
  Scale (Never; Sometimes; Often; Always)
Making Social Connections (New or Reestablished) | Baseline, Session 2 [Experimental Condition Only], Immediate Follow-Up (3 Weeks), 3 months, 6 months
  Measures:
  How many new social connections were established (since the beginning of the study)?
  How many old social connections were re-established (since the beginning of the study)?
  Continuous (Numeric)

OTHER OUTCOMES:
Seeking Substance Use or Mental Health Treatment or Recovery Services | Baseline, Session 2 [Experimental Condition Only], Immediate Follow-Up (3 Weeks), 3 months, 6 months
  Measures:
  See a mental health professional if there concerns or substance use Attend a 12-step group if previous substance use Attend another abstinence-based program if previous substance use Attend a substance use treatment program that uses medications if previous substance use Attend a faith-based substance use group
  Binary (Yes/No)
  Research team reported referrals provided to participants healthcare and mental health/substance use recovery.
  Continuous (Numeric)
Interacting Positively with People Who Use Substances During and Outside the Sessions and Drug Stigma | Baseline, Session 2 [Experimental Condition Only], Immediate Follow-Up (3 Weeks), 3 months, 6 months
  Measures:
  The following items will be combined into a composite measure of drug stigma.
  Refrain from using hurtful language to refer to people with substance use disorder, Refrain from using hurtful language to refer to people from other groups (e.g., religious), Intend to say something to intervene when someone uses hurtful language
  Scale (Never; Sometimes; Almost Always; Always)
  People who use drugs are to blame for their drug use, People who use drugs are dangerous, People who use drugs should be excluded from society, People with a mental health condition are to blame for their condition, People with a mental health condition are dangerous, People with a mental health condition should be excluded from society.
  Scale (Strongly disagree; somewhat disagree; neither disagree not agree; somewhat agree; strongly agree)
Substance Use Without a Prescription or More Than Prescribed (With Baseline Level at 3 and 6 Months) | Baseline, Session 2 [Experimental Condition Only], Immediate Follow-Up (3 Weeks), 3 months, 6 months
  Measures:
  Use substance without a prescription or more than prescribed, Drink alcohol frequency
  Scale (Never; A few times but not in the past year Once a month; A few times a month Once a week; A few times a week Once a day; More than once a day)
Injection Substance Use (With Baseline Level at 3 and 6 Months) | Baseline, Session 2 [Experimental Condition Only], Immediate Follow-Up (3 Weeks), 3 months, 6 months
  Measures:
  Inject substances
  Scale (Never; A few times but not in the past year Once a month; A few times a month Once a week; A few times a week Once a day; More than once a day)
Seeking Treatment for HIV and HCV if Participant is Seropositive | Baseline, Session 2 [Experimental Condition Only], Immediate Follow-Up (3 Weeks), 3 months, 6 months
  Measures:
  Seeking treatment for HIV/HCV if they test positive
  Binary (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Albarracin, PhD, Principal Investigator — Univ. of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT05363865/SAP_000.pdf